CLINICAL TRIAL: NCT00963547
Title: A Phase I Investigation of the Combination of MK-2206, Trastuzumab and Lapatinib in HER2+ Solid Tumors
Brief Title: A Study of MK-2206 in Combination With Trastuzumab and Lapatinib for the Treatment of HER2+ Solid Tumors (MK-2206-015)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2206-015; 2009_646; MK-2206-015 (Other: Merck Protocol Number); 2009-012661-59 (EudraCT Number)
Record Dates: First submitted 2009-08-19; First posted 2009-08-21 (Estimated); Results first posted 2018-10-31 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Advanced Solid Tumors; Breast Cancer
Keywords: Documented to be HER2+
MeSH Terms: conditions — Breast Neoplasms | interventions — MK 2206; Trastuzumab; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Pt. 1: MK-2206 45mg, QOD + Trastuzumab (Experimental): Participants in Part 1 (Pt. 1) receive MK-2206 45 mg every other day (QOD), taken orally. In combination with MK-2206, trastuzumab is administered by intravenous (IV) infusion at an initial dose of 8 mg/kg (loading dose) followed by 6 mg/kg every 3 weeks (q3wk).
  Interventions: Drug: MK-2206; Biological: Trastuzumab
- Pt. 1: MK-2206 60mg, QOD + Trastuzumab (Experimental): Participants in Pt. 1 receive MK-2206 60 mg QOD, taken orally. In combination with MK-2206, trastuzumab is administered by IV infusion at an initial dose of 8 mg/kg (loading dose) followed by 6 mg/kg q3wk.
  Interventions: Drug: MK-2206; Biological: Trastuzumab
- Pt. 1: MK-2206 135mg, QW + Trastuzumab (Experimental): Participants in Pt. 1 receive MK-2206 135 mg once weekly (QW), taken orally. In combination with MK-2206, trastuzumab is administered by IV infusion at an initial dose of 8 mg/kg (loading dose) followed by 6 mg/kg q3wk.
  Interventions: Drug: MK-2206; Biological: Trastuzumab
- Pt. 1: MK-2206 200mg, QW + Trastuzumab (Experimental): Participants in Pt. 1 receive MK-2206 200 mg QW, taken orally. In combination with MK-2206, trastuzumab is administered by IV infusion at an initial dose of 8 mg/kg (loading dose) followed by 6 mg/kg q3wk.
  Interventions: Drug: MK-2206; Biological: Trastuzumab
- Pt. 2: MK-2206 (Pt.1 MTD) + Trastuzumab + Lapatinib 500mg, QD (Experimental): Participants in Part 2 (Pt. 2) receive MK-2206 (dosed either QOD or QW) taken orally at the maximum tolerated dose defined in Part 1 (Pt. 1 MTD). MK-2206 is administered in combination with trastuzumab (IV infusion at an initial dose of 8 mg/kg (loading dose) followed by 6 mg/kg q3wk) as well as lapatinib 500 mg taken orally once daily (QD).
  Interventions: Drug: MK-2206; Biological: Trastuzumab; Drug: Lapatinib
- Pt. 2: MK-2206 (Pt.1 MTD) + Trastuzumab + Lapatinib 750mg, QD (Experimental): Participants in Pt. 2 receive MK-2206 (dosed either QOD or QW) taken orally at the Pt. 1 MTD. MK-2206 is administered in combination with trastuzumab (IV infusion at an initial dose of 8 mg/kg (loading dose) followed by 6 mg/kg q3wk) as well as lapatinib 750 mg taken orally QD.
  Interventions: Drug: MK-2206; Biological: Trastuzumab; Drug: Lapatinib
- Pt. 2: MK-2206 (Pt.1 MTD) + Trastuzumab + Lapatinib 1000mg, QD (Experimental): Participants in Part 2 (Pt. 2) receive MK-2206 (dosed either QOD or QW) taken orally at the Pt. 1 MTD. MK-2206 is administered in combination with trastuzumab (IV infusion at an initial dose of 8 mg/kg (loading dose) followed by 6 mg/kg q3wk) as well as lapatinib 1000 mg taken orally QD.
  Interventions: Drug: MK-2206; Biological: Trastuzumab; Drug: Lapatinib

INTERVENTIONS:
Drug: MK-2206 — [Part 1]: MK-2206 tablets will be given starting at a dose of 45 mg QOD and escalated to 60 mg QOD if tolerated, OR starting at a dose of 135 mg QW and escalated to 200 mg QW if tolerated. Dose reduction to 30mg QOD or 90 mg QW may be permitted. The dose of MK2206 will be increased or decreased as required to find the maximum tolerated dose (MTD) of MK2206 for both the QOD and QW dosing schedules in combination with trastuzumab. [Part 2] The Part 2 dosing level and schedule of MK2206 will be chosen from the MTD of either the QOD or QW dosing schedules depending on the toxicity profile and preliminary efficacy.
Biological: Trastuzumab — Trastuzumab will be administered as a 90-minute IV infusion at a loading dose of 8 mg/kg followed by 6 mg/kg q3wk.
Drug: Lapatinib — Lapatinib tablets will be administered orally QD in doses of 500 mg, 750 mg, or 1000 mg.
  Arms: Pt. 2: MK-2206 (Pt.1 MTD) + Trastuzumab + Lapatinib 1000mg, QD; Pt. 2: MK-2206 (Pt.1 MTD) + Trastuzumab + Lapatinib 500mg, QD; Pt. 2: MK-2206 (Pt.1 MTD) + Trastuzumab + Lapatinib 750mg, QD

SUMMARY:
This study will assess the safety, tolerability, and the maximum tolerated dose (MTD) of MK-2206 in combination with both trastuzumab and trastuzumab/lapatinib in participants with human epidermal growth factor receptor 2 positive (HER2+) breast cancer and other solid tumors. The primary hypothesis of this study is that the combination of oral MK-2206 with trastuzumab or with trastuzumab/lapatinib will be well tolerated in participants with advanced HER2+ solid tumors.

DETAILED DESCRIPTION:
This study was divided into 2 parts. In Part 1, cohorts of 3 participants were to be enrolled sequentially on escalating doses of MK-2206 in combination with a fixed dose of trastuzumab. Barring dose-limiting toxicities (DLTs), additional participants were to be enrolled and dose-finding would proceed until an MTD was identified for MK-2206 when dosed either every other day (QOD) or once weekly (QW) in combination with trastuzumab. In Part 2, cohorts of 3 participants were to be enrolled sequentially on rising doses of lapatinib administered in combination with the MTD dose of MK-2206/trastuzumab established in Part 1. Barring DLTs, dose finding would proceed until an MTD of the 3-drug combination was identified.

ELIGIBILITY:
Inclusion Criteria:

* Have a histologically or cytologically-confirmed locally advanced or metastatic HER2+ solid tumor.
* Have performance status ≤1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Have adequate organ function.
* Female participants have a negative pregnancy test 72 hours prior to receiving the first dose of study medication.
* Have completed any major surgery for a minimum of 28 days prior to enrollment in this study.
* Able to swallow tablets and has no surgical or anatomical condition that will preclude the patient from swallowing or absorbing oral medications on an ongoing basis.

Exclusion Criteria:

* Had chemotherapy, radiotherapy or biological therapy within 4 weeks of screening. Participants receiving trastuzumab and/or lapatinib prior to screening must be off both medications for 1 week prior to first dose of MK-2206 if trastuzumab had been administered at 2 mg/kg weekly and 3 weeks if trastuzumab had been administered at 6 mg/kg weekly.
* Currently participating or has participated in a study with an investigational compound or device within 30 days, or 5x half-life from prior agents, whichever is longer, of Day 1 of this study
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has a primary CNS tumor.
* Has known hypersensitivity to the components of study drugs or its analogs.
* Has a history or evidence of heart disease.
* Has uncontrolled hypertension or diabetes.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding or is expecting to conceive or father children during the study.
* Is HIV positive.
* Has symptomatic ascites or pleural effusion.
* Is receiving treatment with oral corticosteroids for reason other than CNS metastasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-09-15 (Actual); Primary Completion 2011-08-09 (Actual); Study Completion 2011-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Hudis C, Swanton C, Janjigian YY, Lee R, Sutherland S, Lehman R, Chandarlapaty S, Hamilton N, Gajria D, Knowles J, Shah J, Shannon K, Tetteh E, Sullivan DM, Moreno C, Yan L, Han HS. A phase 1 study evaluating the combination of an allosteric AKT inhibitor (MK-2206) and trastuzumab in patients with HER2-positive solid tumors. Breast Cancer Res. 2013 Nov 19;15(6):R110. doi: 10.1186/bcr3577. PMID 24252402

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Per protocol, this trial was to be conducted in 2 parts. In Part 1 (Pt. 1), 33 participants were enrolled, with 31 participants receiving study treatment. Due to trial termination, enrollment into the study was discontinued and Part 2 (Pt. 2) did not begin.
Groups:
- Pt. 2: MK-2206 (Pt.1 MTD) + Trastuzumab + Lapatinib 1000mg, QD: Participants in Pt. 2 receive MK-2206 (dosed either QOD or QW) taken orally at the Pt. 1 MTD. MK-2206 is administered in combination with trastuzumab (IV infusion at an initial dose of 8 mg/kg (loading dose) followed by 6 mg/kg q3wk) as well as lapatinib 1000 mg taken orally QD.
Period: Overall Study
Arm/Group | Pt. 1: MK-2206 45mg, QOD + Trastuzumab | Pt. 1: MK-2206 60mg, QOD + Trastuzumab | Pt. 1: MK-2206 135mg, QW + Trastuzumab | Pt. 1: MK-2206 200mg, QW + Trastuzumab | Pt. 2: MK-2206 (Pt.1 MTD) + Trastuzumab + Lapatinib 500mg, QD | Pt. 2: MK-2206 (Pt.1 MTD) + Trastuzumab + Lapatinib 750mg, QD | Pt. 2: MK-2206 (Pt.1 MTD) + Trastuzumab + Lapatinib 1000mg, QD
Started | 4 | 11 | 12 | 6 | 0 (Study terminated before Part 2 enrollment.) | 0 (Study terminated before Part 2 enrollment.) | 0 (Study terminated before Part 2 enrollment.)
Treated | 3 | 11 | 11 | 6 | 0 (Study terminated before Part 2 enrollment.) | 0 (Study terminated before Part 2 enrollment.) | 0 (Study terminated before Part 2 enrollment.)
Completed | 0 | 0 | 0 | 0 | 0 (Study terminated before Part 2 enrollment.) | 0 (Study terminated before Part 2 enrollment.) | 0 (Study terminated before Part 2 enrollment.)
Not Completed | 4 | 11 | 12 | 6 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 3 | 8 | 9 | 5 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Reason Unknown | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population includes all participants receiving ≥1 dose of study treatment.
Groups:
- Pt. 1: MK-2206 45mg, QOD + Trastuzumab: Participants in Pt. 1 receive MK-2206 45 mg QOD, taken orally. In combination with MK-2206, trastuzumab is administered by IV infusion at an initial dose of 8 mg/kg (loading dose) followed by 6 mg/kg q3wk.
- Pt. 1: MK-2206 135mg, QW + Trastuzumab: Participants in Pt. 1 receive MK-2206 135 mg QW, taken orally. In combination with MK-2206, trastuzumab is administered by IV infusion at an initial dose of 8 mg/kg (loading dose) followed by 6 mg/kg q3wk.
- Total: Total of all reporting groups
Arm/Group | Pt. 1: MK-2206 45mg, QOD + Trastuzumab | Pt. 1: MK-2206 60mg, QOD + Trastuzumab | Pt. 1: MK-2206 135mg, QW + Trastuzumab | Pt. 1: MK-2206 200mg, QW + Trastuzumab | Total
Number analyzed (Participants) | 3 | 11 | 11 | 6 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.0 (8.2) | 55.2 (6.9) | 49.6 (7.4) | 49.7 (7.4) | 51.2 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 10 | 11 | 4 | 28
  Male | 0 | 1 | 0 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing ≥1 Adverse Event
Description: The number of participants experiencing an adverse event (AE) was assessed. An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the sponsor's product, whether or not considered related to the use of the product. Further, any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the sponsor's product, is also an AE.
Time Frame: Up to 36 weeks (up to 4 weeks following cessation of study treatment)
Population: All participants in Part 1 receiving ≥1 dose of study medication (i.e. all participants as treated). Due to trial termination, participants were not enrolled in Part 2; Part 2-specific arms are not included for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Pt. 1: MK-2206 45mg, QOD + Trastuzumab | Pt. 1: MK-2206 60mg, QOD + Trastuzumab | Pt. 1: MK-2206 135mg, QW + Trastuzumab | Pt. 1: MK-2206 200mg, QW + Trastuzumab
Number analyzed (Participants) | 3 | 11 | 11 | 6
Participants | 3 | 11 | 11 | 6

2. Primary Outcome: Number of Participants Discontinuing Study Drug Due to an Adverse Event
Description: The number of participants discontinuing study drug due to an AE was assessed. An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the sponsor's product, whether or not considered related to the use of the product. Further, any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the sponsor's product, is also an AE.
Time Frame: Up to 32 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pt. 1: MK-2206 45mg, QOD + Trastuzumab | Pt. 1: MK-2206 60mg, QOD + Trastuzumab | Pt. 1: MK-2206 135mg, QW + Trastuzumab | Pt. 1: MK-2206 200mg, QW + Trastuzumab
Number analyzed (Participants) | 3 | 11 | 11 | 6
Participants | 0 | 1 | 1 | 1

3. Primary Outcome: Number of Participants Experiencing ≥1 Dose-Limiting Toxicity (DLT) in Cycle 1
Description: A DLT is a drug-related AE not related to disease progression or intercurrent illnesses. Toxicities are graded in severity according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCICTCAE) version 3.0. The following are considered DLTs: A.) Hematologic [grade 4 neutropenia (≥5 days); grade 3/4 neutropenia; grade 4 thrombocytopenia.] B.) Non-Hematologic [any grade ≥3 non-hematologic toxicity except: grade 3 nausea, vomiting, diarrhea, or dehydration; asthenia; hypersensitivity; grade 3 elevated transaminases (1 week).] C.) Additional [any drug-related AE leading to MK-2206 dose modification; grade ≥2 drug-related AE causing drug interruption (≥8 days); any drug-related AE causing drug interruption (≥15 days); grade ≥3 glucose intolerance with grade ≥2 hyperglycemia; fasting glucose >250 mg/dL (≥2 days); grade ≥3 electrolyte abnormality; lactoacidosis or ketoacidosis; non-fasting grade 4 hyperglycemia; increased QTc interval; significant bradycardia.].
Time Frame: Up to 3 weeks (up to day 21 of cycle 1)
Population: All participants in Part 1 receiving ≥1 dose of study drug were included: 1) if experiencing a DLT in cycle 1; or 2) if not experiencing a DLT in cycle 1, received 90% of planned doses and completed all safety evaluations by ≤20 days after first dose of MK-2206. Trial terminated before Part 2 enrollment; Part 2-specific arms excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Pt. 1: MK-2206 45mg, QOD + Trastuzumab | Pt. 1: MK-2206 60mg, QOD + Trastuzumab | Pt. 1: MK-2206 135mg, QW + Trastuzumab | Pt. 1: MK-2206 200mg, QW + Trastuzumab
Number analyzed (Participants) | 3 | 11 | 11 | 6
Participants | 0 | 1 | 1 | 2

4. Primary Outcome: Maximum Tolerated Dose of MK-2206 in Combination With Trastuzumab (Part 1) and With Trastuzumab/Lapatinib (Part 2)
Description: The maximum tolerated dose (MTD) of MK-2206 in combination with trastuzumab (Part 1) was assessed for both QOD and QW dosing schedules. To calculate MTD, a dose-response curve for the rate of patients in each treatment combination arm experiencing a DLT in Cycle 1 will be estimated using the pooling-of-adjacent-violators algorithm, with this dose-response curve used to determine the MTD. The MTD is defined as the dose at which the percentage of patients experiencing a DLT is the closest to 25% or 30% in Part 1 and Part 2, respectively. As the study was terminated prior to Part 2 enrollment, the MTD of MK-2206 in combination with trastuzumab/lapatinib could not be determined.
Time Frame: Up to 3 weeks (up to day 21 of cycle 1)
Population: All participants in Part 1 receiving ≥1 dose of study medication (i.e. all participants as treated), categorized by QOD or QW dosing of MK-2206. Due to trial termination, participants were not enrolled in Part 2; MTD could not be calculated for Part 2.
Measure: Number; unit: mg
Groups:
- Pt. 1: MK-2206 (QOD Dosing) + Trastuzumab: Participants in Pt. 1 receive MK-2206 (at 45 or 60 mg) QOD, taken orally. In combination with MK-2206, trastuzumab is administered by IV infusion at an initial dose of 8 mg/kg (loading dose) followed by 6 mg/kg q3wk.
- Pt. 1: MK-2206 (QW Dosing) + Trastuzumab: Participants in Pt. 1 receive MK-2206 (135 or 200 mg) QW, taken orally. In combination with MK-2206, trastuzumab is administered by IV infusion at an initial dose of 8 mg/kg (loading dose) followed by 6 mg/kg q3wk.
- Pt. 2: MK-2206 (Pt.1 MTD) + Trastuzumab + Lapatinib: Participants in Pt. 2 receive MK-2206 (dosed either QOD or QW) taken orally at the Pt. 1 MTD. MK-2206 is administered in combination with trastuzumab (IV infusion at an initial dose of 8 mg/kg (loading dose) followed by 6 mg/kg q3wk) as well as lapatinib at 500, 750, or 1000 mg taken orally QD.
Arm/Group | Pt. 1: MK-2206 (QOD Dosing) + Trastuzumab | Pt. 1: MK-2206 (QW Dosing) + Trastuzumab | Pt. 2: MK-2206 (Pt.1 MTD) + Trastuzumab + Lapatinib
Number analyzed (Participants) | 14 | 17 | 0
mg | 60 | 200 |

5. Primary Outcome: Recommended Phase 2 Dose of MK-2206 in Combination With Trastuzumab (Part 1) and With Trastuzumab/Lapatinib (Part 2)
Description: The recommended phase 2 dose (RP2D) of MK-2206 in combination with trastuzumab (Part 1) was assessed. Data from Part 1 informing the determination of the MTD (i.e. DLTs in cycle 1), along with safety and tolerability data, and the pharmacokinetic profile was used to determine the RP2D for both the QOD and QW dosing of MK-2206 in combination with trastuzumab. As the study was terminated prior to Part 2 enrollment, the RP2D of MK-2206 in combination with trastuzumab/lapatinib could not be determined.
Time Frame: Up to 36 weeks (up to 4 weeks following cessation of study treatment)
Population: All participants in Part 1 receiving ≥1 dose of study medication (i.e. all participants as treated), categorized by QOD or QW dosing of MK-2206. Due to trial termination, participants were not enrolled in Part 2; RP2D could not be calculated for Part 2.
Measure: Number; unit: mg
Arm/Group | Pt. 1: MK-2206 (QOD Dosing) + Trastuzumab | Pt. 1: MK-2206 (QW Dosing) + Trastuzumab | Pt. 2: MK-2206 (Pt.1 MTD) + Trastuzumab + Lapatinib
Number analyzed (Participants) | 14 | 17 | 0
mg | 60 | 135 |

ADVERSE EVENTS:
Time Frame: Up to 36 weeks (up to 4 weeks following cessation of study treatment)
Description: All participants in Part 1 receiving ≥1 dose of study medication (i.e. all participants as treated). Due to trial termination, participants were not enrolled in Part 2; AEs were not collected for Part 2-specific arms.
Arm/Group | Pt. 1: MK-2206 45mg, QOD + Trastuzumab | Pt. 1: MK-2206 60mg, QOD + Trastuzumab | Pt. 1: MK-2206 135mg, QW + Trastuzumab | Pt. 1: MK-2206 200mg, QW + Trastuzumab
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/11 | 0/11 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 5/11 | 5/11 | 3/6
Other Adverse Events (participants affected / at risk) | 3/3 | 11/11 | 11/11 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pt. 1: MK-2206 45mg, QOD + Trastuzumab (N=3) | Pt. 1: MK-2206 60mg, QOD + Trastuzumab (N=11) | Pt. 1: MK-2206 135mg, QW + Trastuzumab (N=11) | Pt. 1: MK-2206 200mg, QW + Trastuzumab (N=6)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic mass (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pt. 1: MK-2206 45mg, QOD + Trastuzumab (N=3) | Pt. 1: MK-2206 60mg, QOD + Trastuzumab (N=11) | Pt. 1: MK-2206 135mg, QW + Trastuzumab (N=11) | Pt. 1: MK-2206 200mg, QW + Trastuzumab (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (4) | 3 (3) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 1 (2) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal tear (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cheilosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (4) | 4 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (4) | 5 (5) | 4 (7) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (5) | 4 (6) | 5 (7) | 3 (3)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal tenesmus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 4 (4) | 1 (3)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (6) | 4 (4) | 2 (4) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 9 (10) | 6 (11) | 5 (6)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (4)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incision site complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 3 (3) | 4 (8)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 3 (3) | 3 (5) | 5 (8)
Blood albumin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 4 (4) | 5 (7) | 4 (5)
Blood amylase increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood creatinine increased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood magnesium increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Blood potassium decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 2 (2) | 6 (10) | 2 (4)
International normalised ratio increased (Investigations) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (3) | 1 (2) | 1 (1)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Prothrombin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Red blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
White blood cell count decreased (Investigations) | 0 (0) | 2 (2) | 3 (4) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 7 (7) | 4 (6) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 8 (15) | 4 (4)
Hyperinsulinaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5) | 2 (2) | 1 (1)
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 4 (4) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (3) | 1 (1)
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 2 (3) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 5 (5) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (3) | 2 (2) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 7 (9) | 4 (7) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin fragility (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.